CLINICAL TRIAL: NCT06300307
Title: A Phase 1/2a Double-Blind, Placebo-controlled, Single- and Multiple Ascending Dose Study to Assess the Safety, Tolerability, PK, PD and Efficacy of IV Administration of ATX-01 In Male and Female Participants Aged 18 to 64 With Classic DM1
Brief Title: Study of ATX-01 in Participants With DM1
Acronym: ArthemiR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ARTHEx Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-ATX-01-DM1-1.1
Record Dates: First submitted 2024-02-26; First posted 2024-03-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATX-01 (Experimental): ATX-01 is a formulation of the anti-microRNA 23b (anti-miR-23b), known as X82108, a novel type of antisense oligonucleotide
  Interventions: Drug: ATX-01
- Placebo (Placebo Comparator): Placebo to ATX-01
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATX-01 — Solution for infusion
  Arms: ATX-01
Drug: Placebo — Solution for infusion
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test ATX-01 in participants with myotonic dystrophy type 1 (DM1). The main question it aims to answer is if ATX-01 is safe and well tolerated. The trial will compare the safety and tolerability of ATX-01 and a matching placebo.

There will be a single-ascending dose part of the trial and a multiple-ascending dose part. In the single-ascending dose, participants will receive one dose of ATX-01 or placebo. In the multiple-ascending dose part, participants will receive three doses of ATX-01 or placebo.

ATX-01 is a novel anti-miR (synthetic single stranded oligonucleotide) that inhibits a microRNA called miR-23b.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with a documented clinical diagnosis of DM1 (CTG expansion of >150 repeats in DMPK gene measured in peripheral blood mononuclear cells)
* Ambulatory, defined as able to complete a 10-meter walk/run test at screening without the use of assistive devices such as canes, walkers, or orthoses, except for ankle-foot orthoses
* Presence for >3 seconds of grip myotonia as confirmed by a central reader

Key Exclusion Criteria:

* Participants with congenital DM1
* Medical Research Council Muscle Scale score of less than 4 on ankle dorsiflexion or significant tibialis anterior atrophy that prevents a muscle biopsy
* Use of mexiletine or other agent for myotonia within 21 days or 5 half-lives, whichever is longer, prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 120 days
  To evaluate the safety and tolerability of ATX-01 in adult participants with DM1

SECONDARY OUTCOMES:
Incidence of clinically significant changes in laboratory assessments, electrocardiograms (ECGs), vital signs, suicidal ideation and behavior | Up to 120 days
  To further evaluate the safety and tolerability of ATX-01 in adult participants with DM1
Maximum observed plasma concentration (Cmax) of ATX-01 | Up to 48 hours post-dose
Area under the plasma concentration-time curve (AUC) of ATX-01 | Up to 48 hours post-dose
Video hand opening time | Change from baseline up to 120 days
  To evaluate the efficacy of ATX-01 on myotonia in participants with DM1
Change from baseline in ankle dorsiflexion strength by quantitative myometry | Change from baseline up to 120 days
  To evaluate the effects of ATX-01 in participants with DM1 on ankle dorsiflexion strength
Change from baseline in Impact on Activities of Daily Living questionnaire item scores | Change from baseline up to 120 days
  The Impact on Activities of Daily Living questionnaire is a 7-item patient-reported outcome designed to evaluate the impact of ATX-01 on activities of daily living in participants with DM1.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - UCLA, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of Iowa Health Care - Department of Neurology, Iowa City, Iowa
  - University of Kansas Medical Center, Department of Neurology, Fairway, Kansas
  - Virginia Commonwealth University, Richmond, Virginia
- Centre Intégré Universitaire de Santé et Services Sociaux du Saguenay-Lac-St-Jean, Chicoutimi, Quebec, Canada
- Institute of Myology, Paris, France
- Italy (2):
  - The NeMO Clinical Center in Milan, Neurorehabilitation Unit, University of Milan, Milan
  - Fondazione Policlinico A. Gemelli- IRCCS, Rome
- Radboudumc, Nijmegen, Netherlands
- Hospital Universitario Donostia, Donostia / San Sebastian, Spain
- St. George's University Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided